CLINICAL TRIAL: NCT03386786
Title: Randomized, Controlled Evaluation of Health Partner mHealth for Total Joint Replacement at Penn Medicine Princeton Medical Center
Brief Title: Health Partner Evaluation at Princeton
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to close study due to slow enrollment.
Sponsor: DePuy Orthopaedics (Industry)
Collaborators: Johnson & Johnson Health and Wellness Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSJ_2017_01
Record Dates: First submitted 2017-10-02; First posted 2017-12-29 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Total Knee Arthroplasty; Total Hip Arthroplasty
Keywords: Total Knee Arthroplasty; Total Hip Arthroplasty; Total Knee Replacement; Total Hip Replacement; Hospital Care Plan; mHealth
MeSH Terms: interventions — Telemedicine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Health Partner) (Experimental): The mobile health (mHealth) product, Health Partner for Knees and Hips (Health Partner), is a combination of a mobile application (app) and a web-based portal.
  Interventions: Behavioral: Health Partner
- Control (Other): Patients randomized to Control will receive pre-printed brochures that outline the steps of the care plan for unilateral TKA and THA, as per standard care provided to any unilateral TJA patient receiving care at Princeton Healthcare System (PHCS).
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Health Partner — Health Partner is a combination of a mobile application and a web-based portal.
  Other Names: mHealth
  Arms: Intervention (Health Partner)
Behavioral: Standard Care — Patients randomized to Control will receive pre-printed brochures that outline the steps of the care plan for unilateral TKA and THA, as per standard care provided to any unilateral TJA patient receiving care at Princeton Healthcare System (PHCS).
  Other Names: Control
  Arms: Control

SUMMARY:
This is a prospective, single-center, randomized, comparative, controlled study. Penn Medicine Princeton Medical Center will enroll a total of 296 subjects (18 years or older) who are electing to have total knee or hip replacement surgery. Subjects will be randomized to either the treatment group (Health Partner alongside standard care) or the control group (standard care alone). Health Partner is a combination of a mobile application and a web-based portal. The primary objective is to compare care plan adherence (pre- and post-surgery) for Health Partner vs. control subjects. Secondary objectives include evaluating all-cause medical resource utilization, communication with health care provider, well-being, fear of surgery, confidence in recovery from surgery, sleep, and patient satisfaction for 90 days post-surgery.

ELIGIBILITY:
Subjects meeting all the following specific criteria will be considered for participation in the study:

1. Subject is 18 years or older at the time of consent.
2. Subject must be identified by their provider as needing elective unilateral TKA or THA.
3. Subject must have a valid e-mail address and willing to access their inbox on a regular basis.
4. Subject must possess a smartphone/device capable of downloading the current version of the Health Partner mobile app and be willing to access and use digital materials for this project.
5. Subject must be able to comprehend and comply with the requirements of the study.
6. Subject must be able to speak, read and understand English fluently.
7. Subject is willing to give voluntary, written informed consent to participate in this service evaluation and authorize the transfer of his/her information to the Sponsor and Business Associate.

Subjects will be excluded from participation in the study if they meet any of the following criteria:

1. Subject is not able to follow the standard of care and would require special care or circumstances.
2. Subject scheduled to have TKA or THA less than or equal to 2 weeks (14 days) from the time they are enrolled in the study.
3. Subject is undergoing a revision to a previous surgery.
4. Subject is undergoing TKA or THA following traumatic injury (i.e. fracture).
5. Subject is expected to need another lower limb joint replacement (hip/knee) prior to completing this service evaluation.
6. Subject is a repeat patient and was enrolled in the study previously.
7. Subject has had prior experience with the Health Partner companion app.
8. Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
9. Subject, in the opinion of their healthcare provider, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect his/her ability to complete patient reported questionnaires or be compliant with follow-up requirements.
10. Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
11. Subject has a significant neurological or musculoskeletal disorder(s) or disease that may adversely affect gait or weight bearing activities (e.g., muscular dystrophy, multiple sclerosis, Charcot disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Care Path Behavioral Assessment (CPBA), Pre-surgery | Early post-operative (day after surgery to 6 weeks post-surgery)
  Survey assesses degree of subject adherence with pre-surgical activities
Care Path Behavioral Assessment (CPBA), Post-surgery | Late post-operative (11-13 weeks post-surgery)
  Survey assesses degree of subject adherence with post-surgical activities

SECONDARY OUTCOMES:
Medical Resource Utilization | Late post-operative (11-13 weeks post-surgery)
  Seven questions to evaluate the number and duration of encounters with the healthcare system after surgery
Confidence in Recovery (1-item) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery)
  One question to gauge subject's confidence in their recovery after surgery on a five-point Likert scale
Fear of Surgery (1-item) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to the day before surgery), early post-operative (day after surgery to 6 weeks post-surgery)
  One question to gauge degree to which subject is fearful of surgery on a five-point Likert scale
Adherence (MOS Patient Adherence) | Early post-operative (day after surgery to 6 weeks post-surgery) and late post-operative (11-13 weeks post-surgery)
  The Medical Outcomes Study (MOS) Patient Adherence is a 5-item questionnaire gauging subject self-reported ability to follow doctors' suggestions and the frequency of subject adherence
Well-being (MQLI) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  The Multi-Cultural Quality of Life Index (MQLI) asks respondents to rank ten different areas of their life [self-care and independent functioning, occupational functioning, social-emotional support, community and service support, interpersonal functioning, global perception of quality of life, physical well-being, personal fulfillment, psychological/emotional well-being, and spiritual fulfillment] on a 10-point Likert scale
Well-being (PHCS-WB) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  The Public Health Surveillance Well-Being Scale (PHCS-WB) comprises 10-items gauging self-reported mental, physical, and social components of well-being
Sleep (MOS Sleep Scale) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  The Medical Outcomes Study (MOS) Sleep Scale is a 12-item instrument intended to gauge extent and nature of sleep disturbances
Sleep (2-items) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  Two questions to assess whether subjects had 7-9 hours of restful sleep per night
Communication (STAR-P) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  The STAR-P is a 12-item instrument to gauge subject's perceptions of clinical communication
Communication (1-item) | Baseline (-6 to -3 weeks pre-surgery), pre-operative (-3 weeks to day before surgery), early post-operative (day after surgery to 6 weeks post-surgery), and late post-operative (11-13 weeks post-surgery)
  One question to assess the frequency of subject's communication with their provider

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Puorro, MSN, BN, Principal Investigator — Penn Medicine Princeton Medical Center
Locations (1):
- Penn Medicine Princeton Medical Center, Plainsboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No